CLINICAL TRIAL: NCT06857760
Title: Effects of Three Different Methods Applied to Patients After Spine Surgery on Nausea, Thirst and Comfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Özge İşeri, Assistant Professor, Ondokuz Mayıs University, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A.30.2.ODM.0.20.08/569-677
Record Dates: First submitted 2025-02-22; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Spinal Surgery
Keywords: nausea, thirst, comfort
MeSH Terms: conditions — Nausea | interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): Routine care
- Ice cube (Experimental)
  Interventions: Other: Ice cube
- Mouth wash (Experimental)
  Interventions: Other: Mouth wash
- Menthol lozenge (Experimental)
  Interventions: Other: Menthol lozenge

INTERVENTIONS:
Other: Ice cube — ıce cube
  Arms: Ice cube
Other: Mouth wash — Mouth wash
  Arms: Mouth wash
Other: Menthol lozenge — menthol lozenge
  Arms: Menthol lozenge

SUMMARY:
The aim of this study was to determine the effects of postoperative methods on nausea, thirst and comfort levels of patients undergoing spinal surgery.

DETAILED DESCRIPTION:
Within the scope of this randomized controlled study, it is aimed to evaluate the effectiveness of ice, mouthwash and menthol lozenge interventions to provide effects on postoperative nausea, thirst and comfort in patients undergoing spinal surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent lumbar disc herniation (LDH) surgery
* LDH surgery patients who recieve general anesthesia
* The patients who were conscious
* The duration of surgery is between 0-3 hours

Exclusion Criteria:

* Patients who cannot understand and speak Turkish
* Allergic patients to menthol
* Patients who received spinal anesthesia
* Patients with lesions on the oral mucosa and lips
* Patients requiring intensive care after surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Nausea | once before the application and 60, 120, 180 and 240 min. after arrival at the clinic
  Nausea level: It consists of a numeric scale. Among the numbers, ''0'' corresponds to ''no thirst/nausea'' and ''10'' corresponds to ''very much thirst/nausea''. As the number increases, nausea and thirst will be accepted as increased. There is no cut-off point.
Thirst | once before the application and 60, 120, 180 and 240 min. after arrival at the clinic
  Thirst level: A minimum score of 12 and a maximum score of 60 can be obtained from the scale. The higher the score obtained from the scale, the higher the level of thirst discomfort of the patients.
Comfort | once before the application and 240 min. after arrival at the clinic
  Comfort level: The highest score that can be obtained from the scale is 192 and the lowest score is 48. A high SCS scoring indicates a high comfort level of the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Özge İşeri, PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Amasya Şerefeddin Sabuncuoğlu Hospital, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Since this is a doctoral study, the results can be shared at the end of the thesis